CLINICAL TRIAL: NCT04016844
Title: Transcranial Direct Current Stimulation to Reduce Asymmetric Glucose Uptake in Leg Muscles of Persons With Multiple Sclerosis
Brief Title: tDCS and Glucose Uptake in Leg Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Thorsten Rudroff, Principal Investigator, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201905825
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Scerosis; PET; tDCS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will receive tDCS in one session and SHAM in the other session.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- tDCS first then SHAM effects on glucose uptake in leg muscles (Experimental): tDCS Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time tDCS will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  Sham Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time SHAM will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  Interventions: Device: transcranial direct current stimulation or SHAM

INTERVENTIONS:
Device: transcranial direct current stimulation or SHAM — A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.
  In the sham condition, the participants will receive the initial 30 seconds of stimulation, after which the current will be set to 0. The same tDCS device (Soterix) will be used.

SUMMARY:
This study is to examine the efficacy of tDCS to improving walking in people with Multiple Sclerosis (PwMS).

Our study compromises 1 group of subjects with MS which will attend the lab for three sessions. In the first session, subjects will be consented, complete the Patient Determined Disease Steps (PDDS), the Fatigue Severity Scale (FSS), and maximal voluntary contractions (MVCs) of the right and left knee extensors and flexors to determine the more-affected leg. The second and third sessions will involve whole-body FDG PET imaging. During each of these sessions, the subject will walk for 20 min on a treadmill at a self-selected speed during which time tDCS or SHAM, in a blinded manner, will be applied to the motor cortex (M1) corresponding to the more-affected leg. Approximately 2 minutes into the walking, [18F]fluorodeoxyglucose (FDG) will be administered by IV injection. Immediately after the walking is completed, the subject will be positioned in the PET/CT scanner and a whole body (top of head to toes) PET/CT scan will be acquired for the evaluation of glucose metabolism in the brain, spine, and lower extremities. The third session will be identical to the second session with the exception that the opposite condition (tDCS or SHAM) will be used.

DETAILED DESCRIPTION:
Prospective participants, men and women with MS, will be recruited. The plan is to enroll up to 30 to get 20 evaluable subjects. To accomplish this study, all participants will need to complete 3 sessions. The first session at the INPL and sessions 2 and 3 at PET Imaging Center (0911ZJPP) and the PET Imaging lab in Pappajohn Biomedical Discovery Building. Session 2 and 3 are separated by 5-8 days. The duration of each session will be approximately 120 minutes. We expect data collection to last 6 months.

In the first session, subjects will be consented, complete the PDDS, the Fatigue Severity Scale (FSS), and maximal voluntary contractions (MVCs) of the right and left knee extensors and flexors to determine the more-affected leg. When leg strength difference is less than 10%, the more affected side will be based on self-report. The second and the third sessions will involve 20 min walking on a treadmill at a self-selected speed during which time tDCS or SHAM will be applied to the motor cortex (M1) corresponding to the more-affected leg and [18F]fluorodeoxyglucose will be administered. At the end of the walking period, the subject will be imaged on a PET/CT scanner from top of head to toes.

Prior to sessions 2 and 3, all subjects will be asked to fast (water and medication can be taken during this time) for a minimum of 6 hours prior to the FDG administration. In addition, the blood glucose level will be checked (via Accuchek) prior to FDG administration and the level must be equal to or less than 200 mg/dL in order to proceed with the FDG administration on that day. At the beginning of session 2 and 3, the subject will be weighed and height measured, have a blood glucose level determined via Accuchek as described above, undergo a urine pregnancy test if the subject is of child-bearing potential, and have an IV catheter inserted for FDG administration. The subject will then be moved to the PET Scanner area in Pappajohn Biomedical Discovery Building. The subject will be asked to use the restroom prior to walking on the treadmill. A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCl). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit. The participant will receive tDCS or SHAM throughout the walking (i.e., for 20 min). In the tDCS trial, the intensity will start at 0 mA and will increase to 3 mA over the first 30 seconds. In the sham condition, the participants will receive the initial 30 seconds of stimulation, after which the current will be set to 0.

Two min into the walking test on the treadmill, 10 mCi of [18F]-FDG will be injected IV. Then, the walking test continues until 20 min is reached. When the walking test is completed, the tDCS device will be removed and the subject will be positioned in the PET/CT scanner and a whole body (top of head to toes) PET/CT scan will be acquired.

Ratings of perceived exertion (RPE) will be recorded with the modified Borg 10-point scale (Borg, 1982). The subjects will be instructed to estimate the effort during walking. The scale will be anchored so that 0 denotes the resting state and 10 represents the strongest effort.

No long-term follow-up will be done.

ELIGIBILITY:
Inclusion Criteria:

* medically diagnosed with Multiple Sclerosis (MS)
* 18-70 yrs. of age, moderate disability (Patient Determined Disease Steps (PDDS) core 2-6)
* Self-reported differences in function between legs, able to walk for 20 min.

Exclusion Criteria:

* MS relapse within last 60 days
* inability to fast for 6 hours
* hyperglycemia (fasting blood sugar > 200 mg/dL)
* insulin-dependent diabetes
* high risk for cardiovascular disease (ACSM risk classification)
* changes in disease-modifying medications within last 45 days
* concurrent neurological/neuromuscular disease
* hospitalization within last 90 days
* diagnosed depression
* inability to understand/sign informed consent, pregnant, history of seizure disorders (or on medications known to lower seizure threshold)
* hydrocephalus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 4 Subjects completed active tDCS first and then SHAM.
Pre-assignment Details: All 4 Subjects completed active tDCS first and then SHAM.
Groups:
- tDCS/SHAM Effects on Glucose Uptake in Leg Muscles: tDCS Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time tDCS will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit. Sham Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time SHAM will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  SHAM: In the sham condition, the participants will receive the initial 30 seconds of stimulation, after which the current will be set to 0. The same tDCS device (Soterix) will be used.
Period: Overall Study
Arm/Group | tDCS/SHAM Effects on Glucose Uptake in Leg Muscles
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 4 participants completed tDCS and SHAM.
Arm/Group | tDCS/SHAM Effects on Glucose Uptake in Leg Muscles
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Glucose Uptake in Leg Muscles
Description: Participants are walking on a treadmill with tDCS or SHAM, followed by a positron emission tomography (PET) scan to measure glucose uptake in leg muscles. SUV asymmetry indices (AIs) were calculated to determine the magnitude of asymmetry between the more- and less-affected legs with a previously used equation: ((less-affected side - more-affected side)/((0.5) × (less-affected side + more- affected side)) × 100). An AI value ≥ 10% was considered asymmetric.
Time Frame: Six Months
Measure: Mean (Standard Deviation); unit: Percentage (%)
Groups:
- tDCS Effects on Glucose Uptake in Leg Muscles: tDCS Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time tDCS will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  Transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.
- SHAM Effects on Glucose Uptake in Leg Muscles: SHAM Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time SHAM stimulation will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  SHAM stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.The participants will receive the initial 30 seconds of stimulation, after which the current will be set to 0.
Arm/Group | tDCS Effects on Glucose Uptake in Leg Muscles | SHAM Effects on Glucose Uptake in Leg Muscles
Number analyzed (Participants) | 4 | 4
Percentage (%) | 6.3 (6.2) | 16.4 (13.6)

2. Secondary Outcome: Ratings of Perceived Exertion (RPE)
Description: Ratings of perceived exertion (RPE) will be recorded with the modified Borg 10-point scale (Borg, 1982). The subjects will be instructed to estimate their effort during walking. The scale will be anchored so that 0 denotes the resting state and 10 represents the strongest effort they are able to perform.
Time Frame: Six Months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- tDCS Effects on Glucose Uptake in Leg Muscles: tDCS Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time tDCS will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  Transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.
  Sham Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time SHAM will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  SHAM: In the sham condition, the participants will receive the initial 30 seconds of stimulation, after which the current will be set to 0. The same tDCS device (Soterix) will be used.
- SHAM Effects on Glucose Uptake in Leg Muscles: Sham Block: The subject will walk for 20 min on a treadmill at a self-selected speed during which time SHAM will be applied to the motor cortex (M1) corresponding to the more-affected leg.
  SHAM: Transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit. The participants will receive the initial 30 seconds of stimulation, after which the current will be set to 0.
Arm/Group | tDCS Effects on Glucose Uptake in Leg Muscles | SHAM Effects on Glucose Uptake in Leg Muscles
Number analyzed (Participants) | 4 | 4
units on a scale | 6 (4) | 6 (5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | tDCS/SHAM Effects on Glucose Uptake in Leg Muscles
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04016844/Prot_SAP_001.pdf